CLINICAL TRIAL: NCT02664324
Title: The Multiple Sclerosis Performance Test (MSPT) Device for Functional Assessment of Multiple Sclerosis (MS) Patients
Brief Title: MSPT Device Usability Study
Acronym: MSPT
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 888MS003
Record Dates: First submitted 2015-12-10; First posted 2016-01-27 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this feasibility study is to evaluate the functionality (e.g., as defined by the primary endpoints) of the fully integrated Multiple Sclerosis Performance Test (MSPT) device, when used by unsupervised participants with MS, or related conditions, with a broad range of disability, in multi-clinical-care environments. Secondary objectives include: Participant perception of usability of device; Participant satisfaction with the device; Ascertain the impact of different clinical environments on device usability; Ascertain impact of assistive devices in usability of device; Ascertain functionality of Bluetooth remote as compared with manual timing.

DETAILED DESCRIPTION:
This study does not involve evaluation(s) of the clinical efficacy of the MSPT device or the efficacy of MS therapies. This feasibility study is examining the usability of the fully integrated MSPT device. Study participants will be enrolled for same-day testing.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of MS, or related conditions, such as: Clinically Isolated Syndrome (CIS), Neuromyelitis Optica (NMO), and Transverse Myelitis (TM)
* Literacy of written English language as displayed on software tool
* Ability to understand and comprehend software tool from the audio and visual instructions provided in English

Key Exclusion Criteria:

* Study participants, who in the opinion of the Investigator, have vision impairment that precludes their ability to see the iPad Air2® screen/MSPT device.
* Neurological illnesses/conditions, such as motor or vocal tics (including a diagnosis of Tourette's syndrome), head trauma with significant loss of consciousness (>30 minutes), cerebral palsy, dementia (including mild cognitive impairment and Alzheimer's disease), chronic meningitis, Parkinson's disease, and Huntington's disease.

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patients or patients with related conditions in a clinical care setting.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of study participants successfully completing all modules of the MSPT device | Through study duration (3-4 hours)
  The MSPT software tool builds upon previously validated measures comprising the Multiple Sclerosis Functional Composite (MSFC) that represents a comprehensive functional assessment of MS participants that include: MyHealth: MS -Patient demographic, health and medication information; NeuroQoL - Neurological Quality of Life test -Participant reported; PST Processing Speed Test- Measures mental processing speed; Contrast Sensitivity Test (CST)- 50cm vision test; MDT Manual Dexterity Test- 9 hole peg test; WST Walking Speed Test - Timed 25 foot walk
Percent (%) of study participants successfully completing all modules of the MSPT device | Through study duration (3-4 hours)

SECONDARY OUTCOMES:
Percent (%) of study participants who select agree/strongly agree (questions 1 to 5) or disagree/ strongly disagree (questions 6-9) on appropriate questions on the MSPT Usability Survey | Through study duration (3-4 hours)
  MSPT usability survey is a 10 item paper-based questionnaire to measure participant perception of the usability of the device. A study participant will meet the usability secondary endpoints if usability (agree/strongly agree or disagree/strongly disagree, as appropriate) is selected for 6 or more survey questions.
Percent (%) of study participants who reported being satisfied or completely satisfied with using MSPT device | Through study duration (3-4 hours)
  MSPT satisfaction survey is a 1 item paper-based questionnaire to measure participant satisfaction with the MSPT device.
Difference of manual timed versus Bluetooth timed in Walking Speed Test (WST) as assessed by Timed 25 foot walk | Through study duration (3-4 hours)
  T25FW is a quantitative mobility and leg function performance test where the participant is timed while walking for 25 feet.
The percent (%) of study participants who have usability issues with Bluetooth remote due to use of an assistive device(s) | Through study duration (3-4 hours)
Between-site differences in percent (%) of study participants who select agree/strongly agree (questions 1 to 5) or disagree/ strongly disagree (questions 6 to 9) on appropriate questions on the MSPT Usability Survey | Through study duration (3-4 hours)
Between-site differences in percent (%) of study participants who select satisfied/completely satisfied on MSPT Satisfaction Survey | Through study duration (3-4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (3):
- United States (3):
  - Research Site, Baltimore, Maryland
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio

REFERENCES:
- [Derived] Rhodes JK, Schindler D, Rao SM, Venegas F, Bruzik ET, Gabel W, Williams JR, Phillips GA, Mullen CC, Freiburger JL, Mourany L, Reece C, Miller DM, Bethoux F, Bermel RA, Krupp LB, Mowry EM, Alberts J, Rudick RA. Multiple Sclerosis Performance Test: Technical Development and Usability. Adv Ther. 2019 Jul;36(7):1741-1755. doi: 10.1007/s12325-019-00958-x. Epub 2019 May 3. PMID 31054035